CLINICAL TRIAL: NCT01528371
Title: The Effect of Low Dose of Midazolam on Blood Pressure and Anxiety Scale in White-coat Hypertensive Dental Patients
Brief Title: Effect of Midazolam on White-coat Hypertensive Dental Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okayama University (Other)
Responsible Party: Principal Investigator, Yoshihisa Watanabe, Department of Dental Anesthesiology and Special Care Dentistry,Okayama University Graduate School of Medicine, Dentistry and Pharmaceutical Sciences, Okayama University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: yoshi0112
Record Dates: First submitted 2012-01-23; First posted 2012-02-08 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Transient Hypertension
Keywords: Intravenous sedation; Midazolam; Dental treatment; White-coat hypertension; STAI; Dental patients; Transient hypertension
MeSH Terms: conditions — White Coat Hypertension | interventions — Midazolam; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midazolam (Active Comparator): Intravenous administration of midazolam at dose of 0.02mg/kg
  Interventions: Drug: Midazolam
- NSS (Placebo Comparator): Intravenous administration of saline solution at dose of 0.004ml/kg as a placebo drug
  Interventions: Drug: Normal Saline Solution (NSS)

INTERVENTIONS:
Drug: Midazolam — 1. Investigators select subject from patients for whom the doctor has ordered intravenous sedation. Inclusion criteria is SBP>=140mmHg or DBP>=90mmHg measuring when the patient sits on dental chair and has settled down for 5 minutes. Informed consent is obtained from the patient.
  2. Patient conducts Japanese version of STAI and VAS about anxiety to dental treatment.
  3. Investigators take venous line on the upper limb and inject the drug (midazolam at dose of 0.02mg/kg) intravenously. Investigators measure blood pressure, heart rate, and oxygen saturation every 2 minutes until 10 minutes after drug administration.
  4. 10 minutes later, patient conducts Japanese version of STAI and VAS about anxiety to dental procedure again.
  5. Investigators inject an additional sedative agent and the dental treatment is started.
  Arms: Midazolam
Drug: Normal Saline Solution (NSS) — 1. Investigators select subject from patients for whom the doctor has ordered intravenous sedation. Inclusion criteria is SBP>=140mmHg or DBP>=90mmHg measuring when the patient sits on dental chair and has settled down for 5 minutes. Informed consent is obtained from the patient.
  2. Patient conducts Japanese version of STAI and VAS about anxiety to dental treatment.
  3. Investigators take venous line on the upper limb and inject the drug (saline solution at dose of 0.004ml/kg) intravenously. Investigators measure blood pressure, heart rate, and oxygen saturation every 2 minutes until 10 minutes after drug administration.
  4. 10 minutes later, patient conducts Japanese version of STAI and VAS about anxiety to dental procedure again.
  5. Investigators inject an additional sedative agent and the dental treatment is started.
  Arms: NSS

SUMMARY:
Intravenous sedation was used for dealing with transient hypertension, so-called white-coat hypertension, before dental treatment. Midazolam used as a sedative also has antianxiety effect, and the mechanism is guessed that it minimizes patients' stress, resulting in the stability of blood pressure. The purpose of this randomized controlled trial (RCT) is to evaluate the effect of low dose of midazolam on blood pressure and anxiety scale in white-coat hypertensive dental patients.

ELIGIBILITY:
Inclusion Criteria:

SBP>=140mmHg or DBP>=90mmHg measuring when the patient sits on dental chair and has settled down for 5 minutes among dental outpatients scheduling intravenous sedation with American Society of Anesthesiologists physical status I or II.

Exclusion Criteria:

1. Uncontrolled or unstable hypertension
2. Secondary hypertension such as hyperthyroidism and pheochromocytoma
3. Taking sympathomimetic drugs
4. Contraindication of midazolam such as myasthenia gravis and acute narrow-angle glaucoma
5. A pregnant woman or during lactation period
6. Psychiatric disorder such as schizophrenia
7. Not having intelligence enough to read, understand and write a Japanese version of STAI
8. Judged unsuitable by a researcher

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Until 10 minutes after drug administration
Heart rate | Until 10 minutes after drug administration
Oxygen saturation | Until 10 minutes after drug administration

SECONDARY OUTCOMES:
Visual analog scale about anxiety to dental treatment | 10 minutes after drug administration
Sedation level | 10 minutes after drug administration
Japanese version of STAI | 10 minutes after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihisa Watanabe, DDS, Principal Investigator — Department of Dental Anesthesiology and Special Care Dentistry, Okayama University Graduate School of Medicine, Dentistry and Pharmaceutical Sciences
Locations (1):
- Department of Dental Anesthesiology and Special Care Dentistry, Okayama University Graduate School of Medicine, Dentistry and Pharmaceutical Sciences, Okayama, Japan